CLINICAL TRIAL: NCT00127270
Title: Using Behavioral Therapy in Combination With Drug-Darifenacin for Symptoms of Overactive Bladder
Brief Title: Using Behavioral Therapy in Combination With Darifenacin for Symptoms of Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDAR328AUS01
Record Dates: First submitted 2005-06-30; First posted 2005-08-05 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Urinary Incontinence
Keywords: OAB; Overactive Bladder; Bladder hyperactivity; Urge Incontinence; Incontinence; Bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — darifenacin; Behavior Therapy

ARMS (2):
- 1 (Experimental): Darifenacin
  Interventions: Drug: Darifenacin
- 2 (Other): Darifenacin in combination with Behavioral Modification Programme for Symptoms of Overactive Bladder
  Interventions: Drug: Darifenacin; Behavioral: Behavioral therapy

INTERVENTIONS:
Drug: Darifenacin — Darifenacin tablets 7,5 mg once daily with the possibility to up-titrate to 15 mg once daily
  Other Names: Enablex
  Arms: 1
Drug: Darifenacin — Darifenacin tablets 7,5 mg or 15 mg once daily
  Arms: 2
Behavioral: Behavioral therapy — Behavioral Modification Programme for symptoms of overactive bladder
  Arms: 2

SUMMARY:
This study is designed to investigate the efficacy and safety of treatment of overactive bladder with darifenacin administered alone or in conjunction with behavioral modification therapies.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of overactive bladder
* Capable of independent toileting and completing a micturition diary
* Able to comprehend English and follow study procedures and instructions

Exclusion Criteria:

* Post void residual > 100ml/sec
* Urine flow rate (Qmax) <10ml/sec for males only

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2005-05; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average number of urinations per patient per day at Week 12

SECONDARY OUTCOMES:
Change from baseline in average number of urination episodes per patient per day at Week 2, Week 6
Change from baseline in average number of urge urinary incontinence episodes, urgency episodes, incontinence pads, and nocturnal urinations per day measured at Weeks 2, 6, 12
Quality of Life (baseline, Week 6, Week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corp., Study Director — Novartis Pharmaceutical
Locations (67):
- United States (67):
  - Alabama Research Center, Birmingham, Alabama
  - Quality of Life Medical & Research, Tucson, Arizona
  - UCLA - Urology Sciences Research Foundation, Culver City, California
  - San Diego Center for Urology Care, La Mesa, California
  - Orange County Urology Associates, Laguna Woods, California
  - Atlantic Urology Medical Group, Long Beach, California
  - California Professional Research, Newport Beach, California
  - Private Practice, North Hollywood, California
  - Medical Center for Clinical Research, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Western Clinical Research, Torrance, California
  - Urology Research Options, Aurora, Colorado
  - Western Urologic Associates, Wheat Ridge, Colorado
  - Connecticut Clinical Research Center, Waterbury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Advance Research Institute, New Port Richey, Florida
  - Florida Healthcare Research, Ocala, Florida
  - Winter Park Urology Associates, Orlando, Florida
  - Atlanta Medical Research Institute, Alpharetta, Georgia
  - Shepard Center, Atlanta, Georgia
  - Deerpath Physicians Group, Gurnee, Illinois
  - RMD Clinical Research Institute, Melrose Park, Illinois
  - Southern Illinois Clinical Research Center, O'Fallon, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Urology of Indiana, Indianapolis, Indiana
  - Metropolitan Urology, Jeffersonville, Indiana
  - Urologic Surgery Associates, Overland Park, Kansas
  - Pratt Internal Medicine Group, Pratt, Kansas
  - Cotton-O'Neil Clinic, Topeka, Kansas
  - Hearthland Research Associates, Wichita, Kansas
  - Adult and Pediatric Urology, Saint Cloud, Minnesota
  - Mississippi Urology Clinical Research, Jackson, Mississippi
  - PPS Clinical Research, St Louis, Missouri
  - Washing Univ School of Medicine - Urologic Research Center, St Louis, Missouri
  - Women's Clinic of Lincoln, Lincoln, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Center for Urologic Care, Voorhees Township, New Jersey
  - Central New York Clinical Research, Manlius, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Jacobi Medical Center, The Bronx, New York
  - Northeast Urology Research, Concord, North Carolina
  - Multi Specialty Research Associates of NC, Raleigh, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Private Practice, Edmond, Oklahoma
  - Southern Oregon Health and Wellness, Medford, Oregon
  - Portland Clinic, Portland, Oregon
  - Williamette Women's Health, Tualatin, Oregon
  - Univ. of Pittsburgh Medical Center- Dept of Urology, Pittsburgh, Pennsylvania
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - South Carolina Clinical Research Center, Columbia, South Carolina
  - Doctors for Women, Nashville, Tennessee
  - Medical Arts Clinic, Corsicana, Texas
  - Radiant Research, Dallas, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Advances in Health, Houston, Texas
  - Kelsey Seybold Research Foundation, Houston, Texas
  - R/D Clinical Research, Lake Jackson, Texas
  - Progressive Clinical Research, Centerville, Utah
  - Intermountain Clinical Research, Salt Lake City, Utah
  - Salt Lake Research, Salt Lake City, Utah
  - Virginia Urology, Richmond, Virginia
  - East Coast Clinical Research, Virginia Beach, Virginia
  - Radiant Research, Lakewood, Washington
  - Valley Women's Clinic, Renton, Washington

REFERENCES:
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598